CLINICAL TRIAL: NCT07352800
Title: A Phase 2a Open-label Study to Assess the Safety, Tolerability, and Dosing Regimen of Antithrombotic Heparin Proteoglycan Mimetic APAC in Patients With Peripheral Arterial Occlusive Disease and Chronic Limb-threatening Ischemia Undergoing Endovascular Revascularization
Brief Title: Safety of Antithrombotic Heparin Proteoglycan Mimetic APAC in Peripheral Arterial Occlusive Disease and Chronic Limb-threatening Ischemia
Acronym: HEALING
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aplagon Oy (Industry)
Collaborators: LINK Medical Research AB (Unknown); Estimates OY (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APLA-PAOD-CS02; 2025-522390-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-21; First posted 2026-01-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Arterial Occlusive Disease; Chronic Limb-Threatening Ischemia
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Chronic Limb-Threatening Ischemia | interventions — Heparin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study consists of two Parts - Part A and B, each divided into subparts 1 and 2. In Part A1, patients are randomized (2:1) to APAC and control groups. In Part A2, patients are randomized (2:2:1) to two APAC dose levels and control. In Part B (both subparts B1 and B2), patients will be randomized in 2:1 ratio to APAC and control groups.
Masking Description: Due to the severity of the disease and the planned treatment regimen, blinding is not applicable in order to ensure safety and proper clinical management of patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part A1 (no endovascular procedure) - APAC (Experimental)
  Interventions: Drug: APAC - dose level 0.50 mg/kg,
- Part A1 (no endovascular procedure) - control (Active Comparator)
  Interventions: Other: Unfractionated heparin (UFH)
- Part A2 (no endovascular procedure) - APAC dose level 1 (Experimental)
  Interventions: Drug: APAC dose level 1: 0.25 mg/kg,
- Part A2 (no endovascular procedure) - APAC dose level 2 (Experimental)
  Interventions: Drug: APAC dose level 2: 0.50 mg/kg,
- Part A2 (no endovascular procedure) - vehicle (Other)
  Interventions: Other: Vehicle (sterile saline, NaCL 0.9%)
- Part B1 (endovascular procedure) - APAC (Experimental)
  Interventions: Drug: APAC (single periprocedural dose)
- Part B1 (endovascular procedure) - control (Active Comparator)
  Interventions: Other: Unfractionated heparin (UFH)
- Part B2 (endovascular procedure) - APAC (Experimental)
  Interventions: Drug: APAC
- Part B2 (endovascular procedure) - control (Active Comparator)
  Interventions: Other: Unfractionated heparin (UFH)

INTERVENTIONS:
Drug: APAC - dose level 0.50 mg/kg, — single i.v. dosing
  Arms: Part A1 (no endovascular procedure) - APAC
Other: Unfractionated heparin (UFH) — administered as standard of care
  Arms: Part A1 (no endovascular procedure) - control; Part B1 (endovascular procedure) - control; Part B2 (endovascular procedure) - control
Drug: APAC dose level 1: 0.25 mg/kg, — weekly i.v. dosing for 4 consecutive weeks
  Arms: Part A2 (no endovascular procedure) - APAC dose level 1
Other: Vehicle (sterile saline, NaCL 0.9%) — weekly i.v. dosing for 4 consecutive weeks
  Arms: Part A2 (no endovascular procedure) - vehicle
Drug: APAC dose level 2: 0.50 mg/kg, — weekly i.v. dosing for 4 consecutive weeks
  Arms: Part A2 (no endovascular procedure) - APAC dose level 2
Drug: APAC (single periprocedural dose) — Dose is selected based on Part A data, periprocedural dosing.
  Arms: Part B1 (endovascular procedure) - APAC
Drug: APAC — Dose is selected based on Part A and Part B, periprocedural dosing plus dosing for 4 consecutive weeks.
  Arms: Part B2 (endovascular procedure) - APAC

SUMMARY:
The goal of this study is to learn if a new medicine (called antiplatelet and anticoagulant [APAC]) can help the body to prevent blood clots and whether APAC is safe and well tolerated in patients with blocked or narrowed arteries in their legs (peripheral arterial occlusive disease [PAOD]), and in patients with severely restricted poor blood flow to the legs that threatens limb health (chronic limb-threatening ischemia [CTLI]). The study also aims to find the best dose of the medicine. The study consists of two parts: Part A will include patients with PAOD and CTLI, Part B will only include patients with CTLI who are having a procedure to restore blood flow in their legs. Both parts will be subdivided into two subgroups (A1 and A2, B1 and B2) which will test different APAC doses and compare single dosing to weekly dosing for 4 weeks. APAC is injected into the blood. The possible treatment response will be compared either to a placebo (a look-alike substance that contains no drug), or to the current standard treatment. Patients will participate in the study for up to 90 or 180 days. During this time, patients will be regularly examined and asked to answer questions concerning their quality of life.

DETAILED DESCRIPTION:
Peripheral arterial occlusive disease is a group of vascular disorders characterized by narrowing and occlusion of peripheral arteries, often resulting in gradual reduction of the blood supply to the limbs. The main pathogenic mechanism of PAOD stems from atherosclerosis, thrombo-inflammation and thrombosis (atherothrombosis). Patients with PAOD are at increased risk of major adverse limb events (MALE, defined as above ankle amputation of the index limb or major reintervention) and major adverse cardiovascular events (MACE). The most severe form of PAOD, CTLI, is characterized by severely decreased blood flow to the lower limbs.

This Phase 2a open-label study will evaluate the safety, tolerability, and dosing regimen of the heparin proteoglycan mimetic APAC in patients with PAOD with moderate claudication (Fontaine stage IIa and IIb) and in patients with CLTI (Fontaine stage III and IV) undergoing endovascular revascularization.

The study consists of two parts (Part A and Part B), both with two subparts:

* in Part A1, a single dose will be administered intravenously (i.v.),
* in Part A2, weekly doses will be administered i.v. for 4 weeks,
* in Part B1, a single dose will be administered intra-arterially (i.a) periprocedurally, and
* in Part B2, the first dose will be administered i.a. periprocedurally, followed by weekly i.v. dosing for 4 weeks.

Part A will evaluate APAC in the PAOD/CLTI patient population. The primary objective is to evaluate safety and tolerability of i.v. APAC for single infusion (Part A1) and weekly dosing (Part A2). Secondary objectives include evaluation of the effects of APAC on the clinical status of PAOD, and assessment of pharmacokinetic (PK), pharmacodynamic (PD) and other blood coagulation parameters. In Part A1, patients are randomized (2:1) to APAC and control groups. In Part A2, patients are randomized (2:2:1) to two APAC dose levels and control. In Part A, safety and recommended dose(s) of APAC for Part B are studied. A Safety Review Committee (SRC) will evaluate the Part A1 and Part A2 data after all patients in a group have completed the Day 8 or Day 29 visit, respectively, and decide the use of reserve doses, and recommend the dose(s) for the Part B.

Part B will evaluate APAC in CTLI patients undergoing endovascular revascularization. As primary objective, safety of the selected dose(s) and dosing frequency of periprocedural i.a. and weekly i.v. APAC administration will be evaluated. Secondary objectives aim to establish a dosing regimen (single vs. multiple dosing) and preliminary efficacy. Moreover, PK, PD and other blood coagulation parameters, as well as the effects of APAC on MALE and MACE-free survival and quality of life will be assessed as secondary objectives.

For both subparts (B1 and B2), patients will be randomized in 2:1 ratio to APAC and control groups. Part B1 with periprocedural dosing can start after the favorable SRC statement from Part A1. All other study parts (Part A1 [Day 8], Part A2 [Day 29], and Part B1 [Day 29]) need to be finalized before the start of Part B2.

For all study patients, the duration of screening period is maximum 28 days. Safety and clinical measures will be collected until the end of the follow-up period (Part A1: Day 29, and Parts A2, B1, B2: Day 90). To assess the effects of APAC on clinical outcome and quality of life, study participants will be followed up for 90 days in Part A1 and 180 days in Part A2, Part B1, and Part B2 after the first dose of APAC. The study ends when the patient has completed the Day 90 (Part A1) and Day 180 (Part A2, B1, and B2) telephone survey to assess quality of life.

ELIGIBILITY:
Inclusion Criteria (Parts A1, B1 and B2):

1. Males aged 45-85 years and postmenopausal females (i.e., no menstrual periods for 12 months without an alternative medical cause) up to 85 years.
2. Diagnosed with a. PAOD classification Fontaine stage III or IV , b. the total length of the treatment-targeted arterial segment ≥ 5 cm below the knee lesion(s) based on contrast-enhanced computed tomography angiography (CTA)/magnetic resonance angiography (MRA)/digital subtraction angiography (DSA) (Part B1 and B2), c. superficial forefoot wounds without overt infection and bone invasion (WIfI 0-1 and 2 limited to digits and WIfI infection 0-1) allowed, d. undergoing endovascular intervention. (In Part A1, if prescheduled endovascular intervention would take place before the Day 8 study visit, patient is not to be enrolled.)
3. CTA/MRA/DSA with contrast agent performed within 3 months prior to study enrolment as part of diagnostics of PAOD, with results available in the patient's medical records.
4. Patients should be treated with antithrombotic medication either acetylsalicylic acid (up to 100 mg once a day [QD]) or clopidogrel (up to 75 mg QD) for at least the preceding five days before the first APAC administration.
5. Adequate lipid lowering therapy, as evaluated by the investigator.
6. Capability and willingness to provide valid, voluntary written informed consent for the study.
7. Males must be willing to use a condom and their female partners of childbearing potential (i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile [hysterectomy, bilateral salpingectomy and bilateral oophorectomy]) must be willing to use highly effective contraception while on study treatment. Highly effective methods include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner; and sexual abstinence.
8. Males must refrain from sperm donation while on study treatment.

Inclusion Criteria (Part A2):

1. Males aged 45-85 years and postmenopausal females (i.e., no menstrual periods for 12 months without an alternative medical cause) up to 85 years.
2. Diagnosed with a. PAOD classification Fontaine stage IIa and IIb, b. not prescheduled for endovascular revascularization within 90 days of first APAC administration.
3. Moderate to severe arterial disease, ABI < 0.7.
4. Patients should be capable of performing evaluable treadmill exercise test.
5. Patients should be treated with antithrombotic medication either acetylsalicylic acid (up to 100 mg QD) or clopidogrel (up to 75 mg QD) for at least the preceding five days before the first APAC administration.
6. Adequate lipid lowering therapy, as evaluated by the investigator.
7. Capability and willingness to provide valid, voluntary written informed consent for the study.
8. Males must be willing to use a condom and their female partners of childbearing potential (i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile [hysterectomy, bilateral salpingectomy and bilateral oophorectomy]) must be willing to use highly effective contraception while on study treatment. Highly effective methods include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable); IUD; IUS; bilateral tubal occlusion; vasectomized partner; and sexual abstinence.
9. Males must refrain from sperm donation while on study treatment.

Exclusion Criteria:

1. Any ischemic lesions of the heel and midfoot and lesions (wounds or gangrene) invading bones, joints, or tendons at metatarsophalangeal joints or more proximal sites.
2. Acute limb-threatening ischemia (e.g., thromboembolic disease).
3. Medical history of, or an existing aneurysm.
4. Endovascular revascularization intervention is done from the contralateral side using cross-over access (Part B1 and B2).
5. Medical history of, or condition known to be associated with impaired hemostasis, i.e., increased intracranial bleeding risk e.g., previous history of intracranial hemorrhage, subarachnoidal bleeding, hemorrhagic stroke, thrombotic or thromboembolic stroke, gastrointestinal bleeding within 6 months of enrolment, or retroperitoneal bleeding any time, or any inherited or acquired bleeding disorder, i.e., von Willebrand disease or hemophilia or other relevant diagnosis causing impaired hemostasis.
6. Current use of therapeutic dose of anticoagulation (warfarin, apixaban, rivaroxaban, dabigatran, edoxaban, fondaparinux, or any heparin derivative) for any medical reason. (Use of dual pathway inhibition [= acetylsalicylic acid 100 mg + rivaroxabahn 2.5 mg x 2] is not a contraindication, but will be temporarily halted for the day of intervention and day of repeating dosing)
7. Patients treated with combined antiplatelet agents: aspirin + P2Y12 antagonist (clopidogrel, ticagrelor, prasugrel).
8. Diagnosis of autoimmune diabetes mellitus (Type 1 diabetes, or latent autoimmune diabetes in adults [LADA]) vasculitis, rheumatoid arthritis, inflammatory bowel diseases, or other general autoimmune diseases.
9. Body mass index > 35 kg/m^2.
10. Patients with clinically significant acute infection, as judged by the investigator.
11. Use of non-steroidal anti-inflammatory medications within 2 weeks prior to the first dose of APAC or during the treatment period. If medication for pain is required, paracetamol or tramadol (e.g. an opioid patch) may be used.
12. Use of selective serotonin reuptake inhibitor (SSRI) medication within 2 weeks prior to the first dose of APAC or during the treatment period.
13. Peroral use of glycosaminoglycans or omega 3 or related products within 28 days before IMP treatment.
14. Major surgery, major trauma or any endovascular intervention within the past 90 days or organ biopsy prior to the screening visit or scheduled for such an intervention during the study.
15. Uncontrolled arterial hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg).
16. Blood hemoglobin concentration <120 g/L or > 170 g/L (men) and <110 g/L or >160 g/L (women) at screening.
17. Blood platelet count <150 x 10^9/L or > 450 x10^9/L and/or leukocyte count in the lower reference range or not above >12 x 10^9/L.
18. Clinically significantly prolonged plasma PT (> 1.2-fold) or a value of less than 50% (when normal reference range is 70-130%).
19. APTT above the upper limit of the reference range.
20. Patients with a medical history of heparin-induced thrombocytopenia.
21. Patients with known significant liver disease, incl. an alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) level > 2.5 x the upper limit of normal (ULN) at screening.
22. A diagnosis of severe chronic kidney disease, defined as having an eGFR category 4 or 5 (eGFR < 30 mL/min/1.73 m2 as per calculation of Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) or albuminuria stage A3 (uACR >300 mg/g).
23. Patients with an active malignancy, or who have received treatment for any malignancy including bone marrow transplantation within 5 years before the screening visit, except for localized basal cell or squamous cell skin cancer that has been cured at least 90 days before screening.
24. Previous treatment with APAC.
25. Patients with known allergy or hypersensitivity to heparin, or heparin products, APAC, and/or antiplatelet agents (e.g., aspirin or clopidogrel), and protamine sulphate, the reversal agent for APAC.
26. Participation in an investigational drug or device study within 90 days prior to screening.
27. Patients who have ever received treatment with a gene therapy.
28. Patients with known antiphospholipid antibody syndrome or other known significant thrombophilia (homozygosity for FV Leiden or FIIG20210A mutation, or phospholipid antibody syndrome, deficiency of antithrombin, protein C or protein S or combined thrombophilia).
29. Any concomitant disease or condition or treatment that could interfere with, or the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the patient in this study as judged by the investigator.
30. Patients with severe comorbidities and limited life expectancy as judged by the investigator.
31. Patients unable or unwilling to comply with the protocol or to cooperate fully with the investigator or site personnel.
32. Patients with current and/or history of drug abuse (defined as illicit drug use) or alcohol abuse (defined as daily consumption of more than 23-24 and 12-16 alcoholic drinks per week in males and females, respectively).

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint - Part A: Occurrence and severity of treatment-emergent adverse events (TEAEs) | From baseline to Day 29 (Part A1) and Day 90 (Part A2) after the first dose of APAC
Primary endpoint - Part B: Occurrence and severity of TEAEs | From baseline to Day 90 after the first dose of APAC

SECONDARY OUTCOMES:
Secondary endpoint 1 - Part A: Fontaine classification | Assessed at screening (Day -28 to Day -1), at Day 29, Day 60 (Part A2 only) and Day 90 (Part A2) after the first dose of APAC
  No unit of measure
Secondary endpoint 1 - Part A: Wound Ischemia foot Infection (WIfI) scoring | Assessed at screening (Day -28 to Day -1), at Day 8, Day 15 (Part A2 only), Day 22 (Part A2 only), Day 29, Day 60 (Part A2 only) and Day 90 (Part A2) after the first dose of APAC
  No unit of measure
Secondary endpoint 1 - Part A: Toe-brachial blood pressure index (TBI) and ankle-brachial systolic blood pressure index (ABI) | Assessed at screening (Day -28 to Day -1) at Day 29, Day 60 (Part A2 only) and Day 90 (Part A2) after the first dose of APAC
  No unit of measure
Secondary endpoint 1 - Part A2: Maximal walking distance in a treadmill exercise test | Assessed at screening (Day -28 to Day -1), at Day 29, Day 60 and Day 90 after the first dose of APAC
  Unit of measure: meters
Secondary endpoint 2 - Part A: Changes in PD and PK, and other blood coagulation biomarkers - clotting time, clot formation time and activated clotting time | Assessed at baseline (Day 1), Day 2, Day 8, Day 15 (only Part A2), Day 22 (only Part A2) and Day 29
  Unit of measure: seconds
Secondary endpoint 2 - Part A: Changes in PD and PK, and other blood coagulation biomarkers - Maximum clot firmness | Assessed at baseline (Day 1), Day 2, Day 8, Day 15 (only Part A2), Day 22 (only Part A2) and Day 29
  Unit of measure: millimeter
Secondary endpoint 2 - Part A: Changes in PD and PK and other coagulation parameters - Activated partial thromboplastin time | Assessed at screening (Day -28 to -1), baseline (Day 1), Day 2, Day 8, Day 15 (only Part A2), Day 22 (only Part A2), Day 29, Day 60 (only Part A2) and Day 90 (only Part A2) after the first dose of APAC
  Unit of measure: seconds
Secondary endpoint 2 - Part A: Changes in PD and PK and other coagulation parameters - Anti-Factor IIa activity | Assessed at baseline (Day 1), Day 2, Day 8, Day 15 (only Part A2) and Day 22 (only Part A2) after the first dose of APAC
  Unit of measure: International Units per milliliter (IU/mL)
Secondary endpoint 2 - Part A: Changes in PD and PK and other coagulation parameters - Anti-Factor Xa activity | Assessed at screening (Day -28 to -1), baseline (Day 1), Day 22 (only Part A2), Day 29, Day 60 (only Part A2) and Day 90 (only Part A2) after the first dose of APAC
  Unit of measure: International Units per milliliter (IU/mL)
Secondary endpoint 2 - Part A: Changes in PD and PK and other coagulation parameters - Fibrinogen | Assessed at screening (Day -28 to -1), baseline (Day 1), Day 22 (only Part A2), Day 29, Day 60 (only Part A2) and Day 90 (only Part A2) after the first dose of APAC
  Unit of measure: gram per milliliter (g/mL)
Secondary endpoint 2 - Part A: Changes in PD and PK and other coagulation parameters - von Willebrand factor antigen (VWF:Ag) and von Willebrand factor activity with gain-of function mutant Glycoprotein Ib fragment [VWF:GPIbM]) | Assessed at screening (Day -28 to -1), baseline (Day 1), Day 22 (only Part A2), Day 29, Day 60 (only Part A2) and Day 90 (only Part A2) after the first dose of APAC
  Unit of measure: percent
Secondary endpoint 3 - Part A: Major adverse limb event (MALE)- and major adverse cardiovascular event (MACE)-free survival | Assessed at screening (Day -28 to -1), at Day 29, Day 90 (Part A1) and Day 180 (Part A2) after the first dose of APAC
  Unit of measure: percentage of patients
Secondary endpoint 3 - Part A: Quality of life questionnaire European Quality of life-5 Dimensions-3 Level (EQ-5D-5L) | Assessed at screening (Day -28 to -1), at Day 29, D90 (Part A1) and D180 (Part A2) after the first dose of APAC
  No unit of measure. This questionnaire uses a scale from 0-100 where higher values mean a better outcome.
Secondary endpoint 3 - Part A: Ischemic pain | From screening (Day -28 to -1), at Day 29, D90 (Part A1) and D180 (Part A2) after the first dose of APAC
  Assessed using the visual analog scale ranging from 0-100 where 0 = "No Pain" and 100 = "Worst Pain Imaginable"
Secondary endpoint 3 - Part A: Number of participants with ischemic ulcers or gangrene | From screening (Day -28 to -1), Day 29, D90 (Part A1) and D180 (Part A2) after the first dose of APAC
  No unit of measure. This will be assessed as per the clinicians judgement (Normal/Abnormal, Not clinically significant/Abnormal, Clinically significant).
Secondary endpoint 3 - Part A: Physical performance questionnaire | From screening (Day -28 to -1), at Day 29, D90 (Part A1) and D180 (Part A2) after the first dose of APAC
  No unit of measure.
  This will be assessed by asking participants to report their ability to conduct the following activities: Walking around your home, Walking 1-2 blocks on level ground, Walking 1-2 blocks up a hill, Walking 3-4 blocks on level ground, Hurrying or jogging (as if to catch a bus), Vigorous work or exercise.
  For each activity, participants will be asked to select one of the following answer options: Extremely limited, Quite a bit limited, Moderately limited, Slightly limited, Not at all limited, Limited for other reason or did not do the activity.
Secondary endpoint 1 - Part B: Fontaine classification | Assessed at screening (Day -28 to -1), at Day 29, Day 36, Day 60 and Day 90 after the first dose of APAC
  No unit of measure
Secondary endpoint 1 - Part B: WIfI scoring | Assessed at screening (Day -28 to -1), at Day 8 (only Part B2), Day 15 (only Part B2), Day 29, Day 36, Day 60 and Day 90 after the first dose of APAC
  No unit of measure
Secondary endpoint 1 - Part B: Outcome of recanalization (TBI and ABI) at rest | Assessed at screening (Day -28 to -1), at Day 29, Day 36, Day 60 and Day 90 after the first dose of APAC
  No unit of measure
Secondary endpoint 2 - Part B: Changes in PD and PK, and other blood coagulation biomarkers - Clotting time, clot formation time and activated clotting time | Assessed at baseline (Day 1), Day 2, Day 8, Day 15 (only Part B2), Day 22 (only Part B2), Day 29 and Day 36 (only Part B2)
  Unit of measure: seconds
Secondary endpoint 2 - Part B: Changes in PD and PK, and other blood coagulation biomarkers - Maximum clot firmness | Assessed at baseline (Day 1), Day 2, Day 8, Day 15 (only Part B2), Day 22 (only Part B2), Day 29 and Day 36 (only Part B2)
  Unit of measure: millimeter
Secondary endpoint 2 - Part B: Changes in PD and PK and other coagulation parameters - Activated partial thromboplastin time (APTT) | Assessed at screening (Day -28 to -1), baseline (Day 1), Day 2, Day 8, Day 15 (only Part B2), Day 22 (only Part B2), Day 29, Day 36 (only Part B2), Day 60 (only Part B2) and Day 90 (only Part B2) after the first dose of APAC
  Unit of measure: seconds
Secondary endpoint 2 - Part B: Changes in PD and PK and other coagulation parameters - Anti-Factor IIa activity | Assessed at baseline (Day 1), Day 2, Day 8, Day 15 (only Part A2), Day 22 (only Part A2), and Day 29 after the first dose of APAC
  Unit of measure: International Units per milliliter (IU/mL)
Secondary endpoint 2 - Part B: Changes in PD and PK and other coagulation parameters - Anti-Factor Xa activity | Assessed at screening (Day -28 to -1), baseline (Day 1), Day 29, Day 36 (only Part B2), Day 60 (only Part B2) and Day 90 (only Part B2) after the first dose of APAC
  Unit of measure: International Units per milliliter (IU/mL)
Secondary endpoint 2 - Part B: Changes in PD and PK and other coagulation parameters - Fibrinogen | Assessed at screening (Day -28 to -1), baseline (Day 1), Day 29, Day 36 (only Part B2), Day 60 (only Part B2) and Day 90 (only Part B2) after the first dose of APAC
  Unit of measure: gram per milliliter (g/mL)
Secondary endpoint 2 - Part A: Changes in PD and PK and other coagulation parameters - von Willebrand factor antigen (VWF:Ag) and von Willebrand factor activity with gain-of function mutant Glycoprotein Ib fragment (VWF:GPIbM)) | Assessed at screening (Day -28 to -1), baseline (Day 1), Day 29, Day 36 (Part B2), Day 60 (only Part B2) and Day 90 (only Part B2) after the first dose of APAC
  Unit of measure: percent
Secondary endpoint 3 - Part B: MALE and MACE-free survival | Assessed at screening (Day -28 to Day -1), at Day 36, Day 90 and Day 180 after the first dose of APAC
  Unit of measure: percentage of patients
Secondary endpoint 3 - Part B: Quality of life questionnaire European Quality of life-5 Dimensions-3 Level (EQ-5D-5L) | Assessed at screening (Day -28 to -1), at Day 36, Day 90 and Day 180 after the first dose of APAC
  No unit of measure. This questionnaire uses a scale from 0-100 where higher values mean a better outcome.
Secondary endpoint 3 - Part B: Ischemic pain | Assessed at screening (Day -28 to -1), at Day 36, Day 90 and Day 180 after the first dose of APAC
  Assessed using the visual analog scale ranging from 0-100 where 0 = "No Pain" and 100 = "Worst Pain Imaginable"
Secondary endpoint 3 - Part B: Number of participants with ischemic ulcers or gangrene | Assessed at screening (Day -28 to -1), at Day 36, Day 90 and Day 180 after the first dose of APAC
  No unit of measure. This will be assessed as per the clinicians judgement (Normal/Abnormal, Not clinically significant/Abnormal, Clinically significant).
Secondary endpoint 3 - Part B: Physical performance questionnaire | Assessed at screening (Day -28 to -1), at Day 36, Day 90 and Day 180 after the first dose of APAC
  No unit of measure.
  This will be assessed by asking participants to report their ability to conduct the following activities: Walking around your home, Walking 1-2 blocks on level ground, Walking 1-2 blocks up a hill, Walking 3-4 blocks on level ground, Hurrying or jogging (as if to catch a bus), Vigorous work or exercise.
  For each activity, participants will be asked to select one of the following answer options: Extremely limited, Quite a bit limited, Moderately limited, Slightly limited, Not at all limited, Limited for other reason or did not do the activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jarna Hannukainen, Study Director — Aplagon Oy
Locations (3):
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No